CLINICAL TRIAL: NCT00757575
Title: Epidemiological Surveillance Network Study To Assess the Disease of Pneumonia in Infants and Children in Japan
Brief Title: Disease Burden of Pneumonia, Meningitis and Bacteremia Among Children in Japan: Pneumonet Japan
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0887X1-4424
Record Dates: First submitted 2008-09-19; First posted 2008-09-23 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Pneumococcal Disease
Keywords: PNEUMONET JAPAN STUDY
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1

SUMMARY:
Streptococcus pneumoniae is a major cause of pneumonia, among infants and children in Japan and worldwideThis study plans to investigate the rate of invasive pneumococcal disease "IPD " and the rate of hospitalizations due to pneumonia in Okinawa and the Eastern half of Hokkaido Currently, only a limited information about pneumococcal disease burden is available in Japan.

ELIGIBILITY:
Eligibility Criteria

- Children residing in the surveillance area(s) aged 28 days to <60 months with clinical suspicion of pneumonia, meningitis and bacteremia who were admitted to the hospital.

Ages: 28 Days to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants and children less than 5 years of age living in Okinawa and Eastern Hokkaido.
Sampling Method: Non-Probability Sample
Enrollment: 28511 (Actual)
Dates: Start 2008-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
1.Describe the distribution of causal pathogen of meningitis and bacteremia 2.Estimate the hospital admission rate of pneumonia patients 3.Estimate the incidence rate of IPD 4.Describe the serotype distribution of S. pneumoniae | 2 years

SECONDARY OUTCOMES:
1.CFRof patients admitted with IPD and/or pneumonia. 2.Antibiotic resistance rate of S. pneumoniae 3.Risk factor distribution 4.Average duration of the hospitalization of patients with IPD, meningitis, and/or pneumonia. | 2-3 years

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (2):
- Japan (2):
  - Kushiro, Hokkaido
  - Naha, Okinawa